CLINICAL TRIAL: NCT02223260
Title: Open-label, Single Dose, Tolerability, Pharmacokinetic/Pharmacodynamics and Safety Study of Dabigatran Etexilate Given at the End of Standard Anticoagulant Therapy in Children Aged Less Than 1 Year Old
Brief Title: Tolerability , PK/PD and Safety of Dabigatran Etexilate Oral Liquid Formulation in Children < 1 Year of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 1160.105; 2014-001259-22 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Results first posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-07

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dabigatran

ARMS (1):
- dabigatran (Experimental): open label arm with dabigatran oral liquid formulation as single dose
  Interventions: Drug: dabigatran

INTERVENTIONS:
Drug: dabigatran — Experimental dose chosen based on age and weight

SUMMARY:
The aim of the study is to investigate the safety and tolerability of dabigatran etexilate solution in children aged less than 1 year, to demonstrate comparable PK/PD relationship to older children and adults and to confirm dabigatran etexilate dosing algorithm for children aged less than 1 year.

DETAILED DESCRIPTION:
Purpose:

ELIGIBILITY:
Inclusion criteria:

* Neonates and infants with aged < 12 months at Visit 1
* Objective diagnosis of VTE
* End of planned treatment course with anticoagulant therapy as per standard of care at the investigator site.
* Written informed consent provided by the patient's parent(s) (or legal guardian) according to local regulations at Visit 1.

Exclusion criteria:

* Weight less than 3 kg at Visit 1
* Conditions associated with an increased risk of bleeding
* renal dysfunction
* hepatic disease
* Anemia or thrombocytopenia at screening

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (4):
- Canada (2):
  - 1160.105.10002 Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - 1160.105.10003 Boehringer Ingelheim Investigational Site, Montreal, Quebec
- 1160.105.33001 Boehringer Ingelheim Investigational Site, Paris, France
- 1160.105.70005 Boehringer Ingelheim Investigational Site, Kazan', Russia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was an open-label, multicentre, multinational, non-randomised, uncontrolled, single dose, single arm Phase IIa study.
Groups:
- Dabigatran Etexilate: The patients were orally administered a single dose of liquid formulation of dabigatran etexilate. The dose were adjusted based on an age and weight (equivalent to a 150 mg dose in adults). In case the patient could not take the full dose at once, the assigned dose could have been given as divided doses.
Period: Overall Study
Arm/Group | Dabigatran Etexilate
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): the treated set included 8 patients who were dispensed study medication and were documented to have taken at least 1 dose of trial medication.
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.912 (1.694)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentrations of Total Dabigatran, 2h and 12 h (+/-2h) Post Administration of Dabigatran Etexilate
Description: Plasma concentrations of total dabigatran, 2h and 12 h (+/-2h) post administration of dabigatran etexilate.
Time Frame: 2 hours (h) and 12h after drug administration on day 1
Population: Pharmacokinetic set (PKS): This patient set included all treated patients who provided at least 1 PK/PD observation and had no important Protocol violations (PVs) with respect to statistical analysis of Pharmacokinetic (PK) or Pharmacodynamic (PD ) endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
ng/mL
  2h | 120.0 (62.1)
  12h | 60.4 (30.0)

2. Primary Outcome: Central Measurement: The Mean aPTT Coagulation Time at 2 h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean activated partial thromboplastin time (aPTT) coagulation time at 2 h and 12 h (±2 h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
Time Frame: 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
second
  E2 | 78.9 (26.7)
  E12 | 62.8 (27.7)

3. Primary Outcome: Central Measurement: The Mean of ECT Coagulation Time at 2 h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean of Ecarin Clotting Time (ECT) coagulation time at 2 h and 12h (+/-2h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
Time Frame: 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
second
  E2 | 101 (44.3)
  E12 | 66.9 (23.5)

4. Primary Outcome: Central Measurement: The Mean of Diluted Thrombin Time (dTT) Coagulation Time at 2 h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean of dTT (AntiFactor IIa activity) coagulation time at 2 h and 12h (+/-2h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
Time Frame: 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
second
  E2 | 48.7 (24)
  E12 | 38.6 (8.12)

5. Primary Outcome: Central Measurement: The Mean aPTT Ratio at 2 h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean aPTT (activated partial thromboplastin time) ratio at 2 h and 12 h (±2 h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
  aPTT ratio= aPTT (post dose)/aPTT (baseline). The mean of aPTT ratio is presented.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
ratio
  ER2 | 1.86 (19.5)
  ER12 | 1.47 (17.7)

6. Primary Outcome: Central Measurement: The Mean ECT Ratio at 2 h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean Ecarin Clotting Time (ECT) ratio at 2 h and 12h (+/-2h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
  ECT ratio= ECT(Post dose)/ECT(baseline), The mean of ECT ratio is presented.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
Ratio
  ER2 | 2.42 (34.2)
  ER12 | 1.63 (13.8)

7. Primary Outcome: Central Measurement: The Mean of dTT Ratio at 2h and 12h (+/-2h) Post Administration of Dabigatran Etexilate.
Description: Central measurement: The mean of dTT (AntiFactor IIa activity) ratio at 2 h and 12 h (±2 h) post administration of dabigatran etexilate. Standard deviation is actually the Coefficient of Variation.
  dTT ratio= dTT(post dose)/dTT(baseline). The mean of dTT ratio is presented.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
ratio
  ER2 | 1.59 (25.4)
  ER12 | 1.26 (5.67)

8. Secondary Outcome: PK-PD Relationship: Relationship Between Total Dabigatran Plasma Concentration and Coagulation Parameters APTT Values.
Description: Linear regression models were used for modeling the relationship between total dabigatran plasma concentration and coagulation parameters APTT values. For our simple regression model, R-squared is equal to the square of Pearson's coefficient of correlation. The R-squared can be between 0 and 1. R-squared =1 means a perfect fit.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Number; unit: R-Square
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
R-Square | 0.752

9. Secondary Outcome: PK-PD Relationship: Relationship Between Total Dabigatran Plasma Concentration and Coagulation Parameters ECT Values.
Description: Linear regression models were used for modeling the relationship between total dabigatran plasma concentration and coagulation parameters ECT values. For our simple regression model, R-squared is equal to the square of Pearson's coefficient of correlation. The R-squared can be between 0 and 1. R-squared =1 means a perfect fit.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Number; unit: R-Square
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
R-Square | 0.858

10. Secondary Outcome: PK-PD Relationship: Relationship Between Total Dabigatran Plasma Concentration and Coagulation Parameters dTT Values.
Description: Linear regression models were used for modeling the relationship between total dabigatran plasma concentration and coagulation parameters dTT (AntiFactor IIa activity) values. For our simple regression model, R-squared is equal to the square of Pearson's coefficient of correlation. The R-squared can be between 0 and 1. R-squared =1 means a perfect fit.
Time Frame: baseline (0.5 h before intake of study medication), 2 h, and 12 h after dosing on day 1
Population: PKS
Measure: Number; unit: R-Square
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
R-Square | 0.920

11. Secondary Outcome: Incidence of All Bleeding Events (Major, CRNM and Minor) During the Treatment Period.
Description: Percentage of patients with Incidence of all bleeding events(major, clinically relevant non-major (CRNM) & minor) during the treatment period (including the residual effect period).Bleeding events were classified as follow:
  Major bleeding: 1) Fatal bleeding 2) Clinically overt bleeding associated with decrease in haemoglobin of at least 2 g/dL (20 g/L) in 24-h-period 3) Bleeding that was retroperitoneal, pulmonary, intracranial, or otherwise involved the central nervous system 4) Bleeding that required surgical intervention in an operating suite. CRNM bleeding: 1) Overt bleeding for which a blood product was administered & which was not directly attributable to the patient's underlying medical condition 2) Bleeding that required medical or surgical intervention to restore haemostasis, other than in an operating suite. Minor bleeding defined as any overt or macroscopic evidence of bleeding that did not fulfil the criteria for either major bleeding or CRNM bleeding.
Time Frame: Within two days after the administration of trial medication, up to 3 days
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
Percentage of participants | 0.0

12. Secondary Outcome: Incidence of All AEs During the Treatment Period
Description: Percentage of patients with all adverse events (AEs) during the treatment period (including REP).
Time Frame: Within two days after the administration of trial medication, up to 3 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
percentage of participants | 0.0

13. Secondary Outcome: Global Assessment of Acceptability and Tolerability of Study Medication
Description: The investigator was to provide a global clinical assessment of tolerability and acceptability of study medication by the patient.This assessment was based on 5-point scale (good, satisfactory, not satisfactory, bad, not assessable).
Time Frame: Day 1 (immediately after dosing)
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Dabigatran Etexilate
Number analyzed (Participants) | 8
percentage of participants
  Good | 75.0
  Satisfactory | 12.5
  Not satisfactory | 0.0
  Bad | 12.5
  Not assessable | 0.0

ADVERSE EVENTS:
Time Frame: Within two days after the administration of trial medication, up to 3 days.
Arm/Group | Dabigatran Etexilate
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.